CLINICAL TRIAL: NCT00132808
Title: A 2-year Randomized, Multicenter, Double-blind, Placebo-controlled Study to Determine the Efficacy and Safety of Intravenous Zoledronic Acid 5 mg Administered Either Annually at Randomization and 12 Months, or Administered at Randomization Only in the Prevention of Bone Loss in Postmenopausal Women With Osteopenia
Brief Title: Zoledronic Acid in the Prevention of Bone Loss in Postmenopausal Women With Osteopenia, 45 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446N2312
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Results first posted 2011-01-10 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Osteopenia
Keywords: Postmenopausal osteoporosis; osteopenia; zoledronic acid; Osteopenia (osteoporosis prevention)
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis, Postmenopausal | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Zoledronic Acid 2x5 mg (Experimental): Zoledronic acid 5 mg intravenous (i.v.) given at randomization and Month 12
  Interventions: Drug: Zoledronic Acid
- Zoledronic Acid 1x5 mg (Experimental): Zoledronic acid 5 mg intravenous (i.v.) given at randomization and placebo at Month 12
  Interventions: Drug: Zoledronic Acid; Drug: Placebo
- Placebo (Placebo Comparator): Placebo given at randomization and Month 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic acid 5 mg intravenous
  Arms: Zoledronic Acid 1x5 mg; Zoledronic Acid 2x5 mg
Drug: Placebo — Physiologic 0.9% normal saline
  Arms: Placebo; Zoledronic Acid 1x5 mg

SUMMARY:
Osteoporosis prevention is important in patients with osteopenia (low bone density). This study will test the safety and efficacy of zoledronic acid in patients diagnosed with osteopenia.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Greater than or equal to 45 years of age
* Osteopenia (lumbar spine bone mineral density [BMD] T-score between -1.0 and -2.5, and BMD T-score > -2.5 at the femoral neck)

Exclusion Criteria:

* Patients with more than one Grade 1 vertebral fracture (as per Genant method; patients with one Grade 1 vertebral fracture are eligible to participate)
* Patients with any Grade 2 or 3 vertebral fracture (as per Genant method)
* Patients with 25-(OH) vitamin D levels less than 15 ng/mL prior to randomization

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2004-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For information regarding facilities, please contact the Central Contact, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Grbic JT, Black DM, Lyles KW, Reid DM, Orwoll E, McClung M, Bucci-Rechtweg C, Su G. The incidence of osteonecrosis of the jaw in patients receiving 5 milligrams of zoledronic acid: data from the health outcomes and reduced incidence with zoledronic acid once yearly clinical trials program. J Am Dent Assoc. 2010 Nov;141(11):1365-70. doi: 10.14219/jada.archive.2010.0082. PMID 21037195
- [Derived] McClung M, Miller P, Recknor C, Mesenbrink P, Bucci-Rechtweg C, Benhamou CL. Zoledronic acid for the prevention of bone loss in postmenopausal women with low bone mass: a randomized controlled trial. Obstet Gynecol. 2009 Nov;114(5):999-1007. doi: 10.1097/AOG.0b013e3181bdce0a. PMID 20168099

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible patients were stratified according to their duration of menopause (those less than 5 years from menopause were included in Stratum I, while those 5 or more years from menopause were included in Stratum II), and randomized equally to one of the three treatment groups.
Groups:
- Zoledronic Acid 1x5 mg: Zoledronic acid 5 mg i.v. given at randomization and placebo at Month 12
Period: Stratum I
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Started | 77 | 70 | 77
Completed | 68 | 58 | 72
Not Completed | 9 | 12 | 5
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lost to Follow-up | 3 | 4 | 1
Not completed — Withdrawal by Subject | 4 | 7 | 3
Not completed — Abnormal test procedure result (s) | 0 | 0 | 1
Period: Stratum II
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Started | 121 | 111 | 125
Completed | 113 | 96 | 116
Not Completed | 8 | 15 | 9
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo | Total
Number analyzed (Participants) | 198 | 181 | 202 | 581
Age, Continuous [Mean (Standard Deviation); unit: years]
  Stratum I (Women < 5 Years From Menopause) | 53.6 (3.62) | 53.7 (3.59) | 54.4 (3.83) | 53.9 (3.68)
  Stratum II (Women >= 5 Years From Menopause) | 63.9 (6.62) | 63.4 (7.74) | 64.2 (7.65) | 63.8 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Data presented for Overall number of Participants and Gender include participants from both strata of the study.
  Participants
    Female | 198 | 181 | 202 | 581
    Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Lumbar Spine Bone Mineral Density (BMD) at Month 24 Relative to Baseline, by Stratum
Description: The percentage change in lumbar spine BMD at Month 24 relative to baseline was derived as 100 x (lumbar spine BMD at 24 Month - lumbar spine BMD at baseline) / (lumbar spine BMD at baseline).
Time Frame: Baseline, Month 24
Population: Intent to treat population. Last observation carried forward (LOCF) was utilized to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Number analyzed (Participants) | 198 | 181 | 202
Percentage change in BMD
  Stratum I (Women < 5 Years From Menopause) | 4.62 (0.444) [5.77 to 7.96] | 4.03 (0.444) [5.15 to 7.39] | -2.24 (0.428) [NA to NA]
  Stratum II (Women >= 5 Years From Menopause) | 5.60 (0.343) [5.32 to 7.17] | 4.76 (0.356) [4.46 to 6.36] | -0.65 (0.339) [NA to NA]

2. Secondary Outcome: Percentage Change in Total Hip BMD at Month 24 Relative to Baseline, by Stratum.
Description: The percentage change in total hip BMD at Month 24 relative to baseline was derived as 100 x (total hip BMD at 24 Month - total hip BMD at baseline) / (total hip BMD at baseline).
Time Frame: Baseline, Month 24
Population: Intent to treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Number analyzed (Participants) | 198 | 181 | 202
Percentage change in BMD
  Stratum I (Women < 5 Years From Menopause) | 2.66 (0.318) [4.00 to 5.52] | 2.55 (0.317) [3.86 to 5.43] | -2.10 (0.293) [NA to NA]
  Stratum II (Women >= 5 Years From Menopause) | 3.04 (0.265) [3.36 to 4.80] | 2.11 (0.282) [2.40 to 3.91] | -1.04 (0.265) [NA to NA]

3. Secondary Outcome: Percentage Change in Femoral Neck BMD at Month 24 Relative to Baseline, by Stratum.
Description: The percentage change in femoral neck BMD at Month 24 relative to baseline was derived as 100 x (femoral neck BMD at 24 Month - femoral neck BMD at baseline) / (femoral neck BMD at baseline).
Time Frame: Baseline, Month 24
Population: Intent to treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Number analyzed (Participants) | 198 | 181 | 202
Percentage change in BMD
  Stratum I (Women < 5 Years From Menopause) | 2.04 (0.550) [2.27 to 4.90] | 2.01 (0.549) [2.20 to 4.92] | -1.55 (0.508) [NA to NA]
  Stratum II (Women >= 5 Years From Menopause) | 2.35 (0.344) [2.60 to 4.47] | 1.46 (0.366) [1.67 to 3.62] | -1.18 (0.343) [NA to NA]

4. Secondary Outcome: Biochemical Marker of Bone Resorption: Serum Beta C-telopeptides (b-CTx), by Stratum
Description: Biomarker: Serum b-CTx levels at Months 6, 12, 18 and 24 by stratum.
Time Frame: Months 6, 12, 18 and 24
Population: Intent to treat population with available data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Number analyzed (Participants) | 198 | 181 | 202
ng/mL
  Stratum I - Month 6 | 0.2217 (0.11791) | 0.2286 (0.09630) | 0.6439 (0.27902)
  Stratum I - Month 12 | 0.2861 (0.13776) | 0.3111 (0.13195) | 0.6634 (0.25433)
  Stratum I - Month 18 | 0.2187 (0.16812) | 0.3605 (0.14847) | 0.6444 (0.28254)
  Stratum I - Month 24 | 0.2864 (0.12242) | 0.3777 (0.14943) | 0.6640 (0.27538)
  Stratum II - Month 6 | 0.1918 (0.12648) | 0.1888 (0.10625) | 0.5802 (0.25034)
  Stratum II - Month 12 | 0.2696 (0.18247) | 0.2484 (0.11435) | 0.5634 (0.23442)
  Stratum II - Month 18 | 0.1986 (0.14900) | 0.2854 (0.14391) | 0.5742 (0.24399)
  Stratum II - Month 24 | 0.2554 (0.17049) | 0.3254 (0.15260) | 0.6012 (0.26942)

5. Secondary Outcome: Biochemical Marker of Bone Formation: Serum N-terminal Propeptide of Type 1 Collagen (P1NP), by Stratum
Description: Biomarker: Serum P1NP levels at Months 6, 12, 18 and 24 by stratum.
Time Frame: Months 6, 12, 18 and 24
Population: Intent to treat population with available data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Number analyzed (Participants) | 198 | 181 | 202
ng/mL
  Stratum I - Month 6 | 20.851 (9.7724) | 20.752 (9.7560) | 59.449 (20.3291)
  Stratum I - Month 12 | 28.231 (12.3748) | 30.500 (14.8217) | 55.166 (20.5274)
  Stratum I - Month 18 | 20.102 (12.6635) | 35.561 (14.1588) | 55.775 (19.8842)
  Stratum I - Month 24 | 28.288 (12.2706) | 38.743 (14.7626) | 56.315 (20.3715)
  Stratum II - Month 6 | 19.369 (14.1819) | 19.423 (16.6028) | 50.271 (22.6624)
  Stratum II - Month 12 | 28.333 (15.8193) | 26.363 (13.1112) | 49.581 (20.6559)
  Stratum II - Month 18 | 19.031 (14.8270) | 29.569 (14.7631) | 46.943 (18.8147)
  Stratum II - Month 24 | 26.211 (11.8566) | 34.418 (15.4474) | 51.621 (20.9281)

6. Secondary Outcome: Biochemical Marker of Bone Formation: Bone Serum Alkaline Phosphatase (BSAP), by Stratum
Description: Biomarker: BSAP levels at Months 6, 12, 18 and 24 by stratum.
Time Frame: Months 6, 12, 18 and 24
Population: Intent to treat population with available data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Number analyzed (Participants) | 198 | 181 | 202
ng/mL
  Stratum I - Month 6 | 8.718 (2.5827) | 8.841 (2.2434) | 13.982 (4.7106)
  Stratum I - Month 12 | 9.945 (2.9027) | 10.539 (2.9800) | 14.127 (4.8981)
  Stratum I - Month 18 | 8.365 (2.5574) | 11.233 (3.1563) | 14.149 (4.8878)
  Stratum I - Month 24 | 9.799 (2.5836) | 11.764 (3.8401) | 14.353 (4.9089)
  Stratum II - Month 6 | 8.219 (2.8126) | 7.925 (2.2847) | 13.394 (5.2169)
  Stratum II - Month 12 | 9.678 (3.0216) | 9.139 (2.4558) | 13.650 (4.8295)
  Stratum II - Month 18 | 8.357 (2.2152) | 10.023 (2.8237) | 13.222 (4.9167)
  Stratum II - Month 24 | 9.730 (2.7591) | 10.916 (3.5878) | 13.902 (4.6302)

ADVERSE EVENTS:
Arm/Group | Zoledronic Acid 2x5 mg | Zoledronic Acid 1x5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 21/198 | 17/181 | 23/202
Other Adverse Events (participants affected / at risk) | 177/198 | 158/181 | 160/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 2x5 mg (N=198) | Zoledronic Acid 1x5 mg (N=181) | Placebo (N=202)
Angina pectoris (Cardiac disorders) | 2 | 1 | 1
Thyroid mass (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 3 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Global amnesia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Endometrial metaplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Leriche syndrome (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 2x5 mg (N=198) | Zoledronic Acid 1x5 mg (N=181) | Placebo (N=202)
Abdominal pain (Gastrointestinal disorders) | 11 | 6 | 6
Constipation (Gastrointestinal disorders) | 13 | 13 | 14
Diarrhoea (Gastrointestinal disorders) | 16 | 12 | 16
Dyspepsia (Gastrointestinal disorders) | 13 | 12 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 5 | 12
Nausea (Gastrointestinal disorders) | 34 | 21 | 16
Vomiting (Gastrointestinal disorders) | 14 | 9 | 9
Asthenia (General disorders) | 12 | 5 | 2
Chills (General disorders) | 36 | 33 | 6
Fatigue (General disorders) | 29 | 18 | 8
Non-cardiac chest pain (General disorders) | 6 | 12 | 6
Oedema peripheral (General disorders) | 11 | 7 | 7
Pain (General disorders) | 48 | 27 | 7
Pyrexia (General disorders) | 43 | 38 | 9
Bronchitis (Infections and infestations) | 12 | 14 | 22
Influenza (Infections and infestations) | 12 | 15 | 12
Nasopharyngitis (Infections and infestations) | 27 | 17 | 23
Sinusitis (Infections and infestations) | 16 | 12 | 24
Upper respiratory tract infection (Infections and infestations) | 27 | 19 | 23
Urinary tract infection (Infections and infestations) | 22 | 16 | 25
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 10 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 | 34 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 30 | 24
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 5 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 10 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 38 | 41 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 12 | 10
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 3 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 29 | 20
Dizziness (Nervous system disorders) | 15 | 11 | 7
Headache (Nervous system disorders) | 29 | 37 | 23
Hypoaesthesia (Nervous system disorders) | 11 | 4 | 3
Insomnia (Psychiatric disorders) | 6 | 5 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 10
Hypertension (Vascular disorders) | 9 | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.